CLINICAL TRIAL: NCT06048419
Title: Acceptability and Efficacy of GO MOVE: A Mobile Health Technology for Youth With Unilateral Cerebral Palsy
Brief Title: Acceptability and Efficacy of GO MOVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Scottish Rite Hospital for Children (Other)
Responsible Party: Principal Investigator, Angela Shierk, Clinical Scientist, Texas Scottish Rite Hospital for Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU-2023-0531
Record Dates: First submitted 2023-08-29; First posted 2023-09-21 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Cerebral Palsy; Hemiplegic Cerebral Palsy
Keywords: home program
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: prospective cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Go Move Home Program (Experimental): Goal driven home program
  Interventions: Behavioral: Home Program

INTERVENTIONS:
Behavioral: Home Program — Home program for 6 weeks (1 hr and 15 minutes per week)

SUMMARY:
The goal of this clinical trial is to learn about the acceptability and efficacy of Go Move, a mobile website developed to assist youth with unilateral cerebral palsy and their caregivers with setting goals and selecting exercises and activities to meet the goals. The main question[s] it aims to answer are:

* Is Go Move accepted by youth with unilateral cerebral palsy and their caregivers?
* Does Go Move support goal attainment for youth with unilateral cerebral palsy?

Participants will set up and participate in a goal-driven home program using the Go Move mobile website. Participants will spend 1 hour and 15 minutes per week for 6 weeks working on their home program and will complete pre-intervention and post-intervention assessments.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for participants to enroll in the study include a diagnosis of unilateral CP or a non-progressive brain lesion, injury, or trauma of the developing brain that presents with a unilateral upper limb motor impairment. GMFCS levels 1 or 2. MACS levels 1-3. Age 3-17 years old, ability to follow directions, ability to complete the assessment protocol, and the ability to access the GO MOVE webpage on a personal device. All ethnic/racial groups will be eligible to participate. The ability to participate in everyday activities without restriction from a physician throughout the duration of their participation in the study (does not have restrictions/contraindications following a medical procedure).

Exclusion Criteria:

* The study will exclude any patients with uncontrolled epilepsy or significant visual impairment. The study will exclude any patient with severe behavioral problems or the inability to complete the assessment protocol or home program.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | within 2 weeks of start of intervention (pre-intervention), within 2 weeks of end of intervention (post-intervention)
  The Canadian Occupational Performance Measure is a criterion referenced, individualized, client-centered outcome measure designed for use by occupational therapists to detect change in a client's self-perception of occupational performance over time on a scale of 1-10 (1 being the lowest)

SECONDARY OUTCOMES:
Goal Attainment Scale (GAS) Light | within 2 weeks of start of intervention (pre-intervention), within 2 weeks of end of intervention (post-intervention)
  The Goal Attainment Scale is an individualized, functional outcome measure involving goal selection and scaling. The scale ranges from -2 to +2 with -2 representing a decline in function, -1 no change, 0 expected outcome, +1 a little more, +2 a lot more.
Assisting Hand Assessment (AHA) (optional) | within 2 weeks of start of intervention (pre-intervention), within 2 weeks of end of intervention (post-intervention)
  The Assisting Hand Assessment is a criterion referenced, valid and reliable 22-item measure that assesses the assisting or affected hand in carrying out bimanual activities for children with cerebral palsy or obstetric brachial plexus palsy measured by AHA units on a scale of 0-100 with 0 being the lowest level of function.

OTHER OUTCOMES:
Demographic information | within 2 weeks of start of intervention (pre-intervention)
  Demographic in formation will be collected including: age in years and months, gender, etiology of cerebral palsy, qualitative description of previous exposure to therapy
Gross Motor Function Classification System (GMFCS) | within 2 weeks of start of intervention (pre-intervention)
  The Gross Motor Function Classification Systems is a 5-level classification system that describes the gross motor function of children and youth with cerebral palsy with 1 being the lowest functioning and 5 being the highest
Manual Ability Classification Scale (MACS) | within 2 weeks of start of intervention (pre-intervention)
  The Manual Ability Classification Scale describes how children with cerebral palsy use their hands during activities of daily living with 1 being the least functional and 5 being the most functional
Mobile App Rating Scale (MARS) | within 2 weeks of end of intervention (post-intervention)
  The Moblie App Rating Scale is an objective, multidimensional tool to assess the quality of mobile health apps using likert scaling with 1 being the lowest rating and 5 being the highest
Feasibility and satisfaction with using the Go Move website | within 2 weeks of end of intervention (post-intervention)
  A likert scale from 1-5 on the satisfaction and ease of using the Go Move website and qualitative data collection with 1 being the lowest rating and 5 being the highest

CONTACTS AND LOCATIONS:
Overall Officials: Angela Shierk, PhD, Principal Investigator — Scottish Rite for Children
Locations (1):
- Scottish Rite for Children, Frisco, Texas, United States

IPD SHARING:
Plan to Share IPD: No